CLINICAL TRIAL: NCT01784341
Title: Circadian Phase in Bipolar Depression: Is it Delayed and Does it Normalize With Remission?
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Gottlieb, Assistant Clinical Professor of Psychiatry, Northwestern University
Other Study IDs: 47709
Record Dates: First submitted 2013-01-29; First posted 2013-02-05 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar, Circadian, Melatonin
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Saliva Samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall aim of this project is to compare sleep patterns and melatonin profiles in individuals with bipolar disorder during depression and after remission. The hypothesis is that sleep time, rest-activity cycles and melatonin onset will be delayed during depression and become less delayed after remission.

DETAILED DESCRIPTION:
Bipolar disorder is a prevalent, disabling, and chronic mood disorder characterized by depressive symptoms that alternate with hypomanic, manic or mixed states. The depressive phase of this illness predominates and is associated with cognitive, occupational and social impairment, psychiatric comorbidity, and increased mortality from suicide and general medical problems. Clarification of the pathophysiology of this illness is important to improve treatment effectiveness.

Various lines of evidence suggest that circadian factors play a role in the onset and maintenance of bipolar depression. Rhythmic clinical disturbances are found in the altered sleep-wake cycle, diurnal mood shifts, rest-activity changes, seasonal features, the cyclic pattern of relapse and remission and the polarity inversions that define this disorder. Chronotherapeutic treatments that act by modifying circadian phase have been shown to be effective in ameliorating the depressive symptoms of this illness. In addition to this circumstantial evidence, there is some more direct data implicating circadian dysfunction in bipolar depression. Genetic studies have documented associations between various circadian genes and bipolar illness. Actigraphic studies of activity levels have demonstrated illness-remission differences and phase advances in manic states. Though these latter studies employ more direct assessment methodologies, there are few articles that have attempted to investigate circadian processes in bipolar depression with the use of the core clock processes. These basic clock rhythms include core body temperature, cortisol levels and dim light melatonin onset. Because these physiological oscillations are less influenced by behavior and less prone to masking, they more accurately reflect the intrinsic timing of the central pacemaker.

This study will use dim light melatonin onset and actigraphy to assess the status and changes in circadian phase between states of bipolar depression and their remission. Using a case control methodology, adult subjects will be evaluated during, and after remission from the depressive phase of bipolar disorder.

General Aim

The overall aim of this project is to compare the timing of dim-light melatonin onset and actigraphy-based activity patterns in adult patients with bipolar disorder in depressed vs remitted states. These markers will enable characterization of changes in circadian phase between illness and recovery. A case control design will enable the use of small sample sizes capable of identifying statistically significant changes in the timing of circadian rhythms in the two states of interest.

Hypotheses

It is predicted that the dim light melatonin onset and activity profile will be delayed in the depressed vs. the euthymic state of bipolar disorder. It is further anticipated that this phase delay will lessen when bipolar subjects achieve remission from their depression.

Last, it is predicted that the circadian phase of the dim light melatonin onset and the activity profile will correlate, both being delayed in the depressive phase, and less delayed in euthymia.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 55
* Bipolar Disorder Type I or II, with current major depression.
* Currently receiving active treatment from a psychiatrist for bipolar disorder

Exclusion Criteria:

* Recent history of, or current Diagnostic and Statistical Manual IV, Text Revision criteria for alcohol or substance abuse/dependence disorders
* circadian rhythm sleep disorders or sleep apnea
* current stimulant use
* any recent or planned transmeridian travel across more than two time zones
* recent, current, or planned shift work schedules
* pregnancy or plan to become pregnant
* a Young Mania Rating Scale Score of greater than or equal to seven
* received in the past two weeks or plan to receive bright light therapy, dawn simulation, sleep deprivation, or other forms of chronotherapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults between 18 and 55 who are currently diagnosed with Bipolar Disorder.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Dim Light Melatonin Onset from Depression to Remission | Collected at end of first and second weeks of actigraphy.
  Subjects will be instructed in the procedures used for home-based, self-collection of saliva samples. The protocol developed by Sit and colleagues at the University of Pittsburgh (attached), will be used. This involves obtaining ten saliva samples, one every 30 minutes, over a 4.5 hour period. This protocol contains instructions about ambient lighting, posture, exercise, eating, and use of the oral swabs and collection kits.

SECONDARY OUTCOMES:
Change in Sleep Schedule from Depression to Remission | One week after initial enrollment and one week after remission of depression.
  Wrist actigraphy and sleep logs will be collected for a one week period to estimate the subjects average sleep schedule.

CONTACTS AND LOCATIONS:
Overall Officials: John Gottlieb, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States